CLINICAL TRIAL: NCT00440518
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of 100mg/Day and 300mg/Day Lacosamide for Migraine Prophylaxis.
Brief Title: A Study Designed to Test the Effectiveness and Safety of Treating Patients With Lacosamide for Migraine Prophylaxis
Acronym: SP906
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SP0906
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Results first posted 2009-09-11 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2017-07

CONDITIONS: Migraine
Keywords: Lacosamide; migraine prophylaxis; Vimpat
MeSH Terms: conditions — Migraine Disorders | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Lacosamide 100mg (Experimental): 100mg lacosamide
  Interventions: Drug: Lacosamide
- Lacosamide 300mg (Experimental): 300mg lacosamide
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide 100mg immediate-release film-coated tablet (white,oval) oral administration twice daily 12 hours apart
  Other Names: LCM; Vimpat
  Arms: Lacosamide 100mg
Other: Placebo — Immediate-release film coated tablet (white, oval), oral administration twice daily 12 hours apart
  Arms: Placebo
Drug: Lacosamide — Lacosamide 300mg, immediate-release film coated tablet (white,oval), oral administration twice daily 12 hours apart.
  Other Names: LCM; Vimpat
  Arms: Lacosamide 300mg

SUMMARY:
The purpose of this study is to see how safe and effective Lacosamide (LCM) is when taken by mouth, twice a day for up to 18 weeks to prevent migraines.

DETAILED DESCRIPTION:
This study is for subjects who have been diagnosed with migraine for at least one year and who are currently taking an effective abortive medication(s).

ELIGIBILITY:
Inclusion Criteria:

* History of migraines headaches for 1 year and well documented 3 month retrospective history of migraines.
* Experience 2-8 migraines per month but not more than 15 headache days per month. There should be at least 48 hours of freedom between headaches.
* On effective stable abortive medication(s) for the acute treatment of migraine.

Exclusion Criteria:

* Subject in another investigational drug or device study within the last 30 days or is currently in another investigational drug trial.
* Use of triptans or ergots for migraine abortive treatment > 2-3 days per calendar week 2 months prior to screening.
* Experience 15 or more headache days per month of any kind 2 months prior to screening.
* Has another consistent or chronic form of headache.
* Unable to stop medications, herbs, vitamins, or minerals used to prevent a migraine from occurring.
* Pregnant or nursing women and those of child bearing potential who are not surgically sterile, or 2 years post menopausal, or do not practice 2 combined methods of birth control, unless sexually abstinent, during the trial.
* Significant laboratory or electrocardiograms (ECG) abnormalities
* Significant medical history including cardiovascular abnormalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (24):
- United States (24):
  - Huntsville, Alabama
  - Little Rock, Arkansas
  - Walnut Creek, California
  - Boulder, Colorado
  - Palm Beach Gardens, Florida
  - South Miami, Florida
  - Sunrise, Florida
  - Conyers, Georgia
  - Evansville, Indiana
  - Wellesley Hills, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Springfield, Missouri
  - St Louis, Missouri
  - Albany, New York
  - Greensboro, North Carolina
  - Matthews, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Alexandria, Virginia
  - Seattle, Washington

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicenter trial with 24 sites with enrolled subjects and 23 sites with randomized subjects from 15 Feb 2007 to 17 Jul 2008.
Pre-assignment Details: Subjects on stable dose of prophylactic medication entered a 2-week Wash-Out Period followed by a 4-week Baseline Period without any prophylactic medication. Subjects not taking prophylactic medication entered the Baseline Period directly for 6 weeks. Subjects entered a 3-week Titration Period and if completed entered a 14-week Maintenance Period.
Groups:
- Placebo: Placebo immediate-release film coated tablet, oral administration twice daily 12 hours apart
- Lacosamide 100mg: Lacosamide 100mg immediate-release film coated tablet, oral administration twice daily 12 hours apart
- Lacosamide 300mg: Lacosamide 300mg immediate-release film coated tablet, oral administration twice daily 12 hours apart
Period: Randomized /Titration Period
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Started | 72 | 72 | 74
Completed | 59 | 63 | 70
Not Completed | 13 | 9 | 4
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Subject Withdrew Consent | 4 | 1 | 0
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Unsatisfactory Compliance | 2 | 3 | 2
Not completed — Other | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Adverse Event | 2 | 3 | 0
Period: Maintenance and Safety Follow-up Periods
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Started | 59 | 63 | 70
Completed | 52 | 51 | 55
Not Completed | 7 | 12 | 15
Not completed — Adverse Event | 3 | 4 | 2
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Subject Withdrew Consent | 3 | 2 | 4
Not completed — Unsatisfactory Compliance | 0 | 3 | 6
Not completed — Other | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg | Total
Number analyzed (Participants) | 72 | 72 | 74 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 72 | 74 | 218
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (12.23) | 40.1 (11.86) | 40.2 (11.40) | 39.9 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 63 | 187
  Male | 10 | 10 | 11 | 31
Region of Enrollment [Number; unit: participants]
  United States | 72 | 72 | 74 | 218

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Migraine Headache Rates During the Entire 14-week Maintenance Period
Time Frame: Baseline, Entire 14-week Maintenance Period
Population: Of the 72 (Placebo), 72 (Lacosamide 100mg) and 74 (Lacosamide 300mg) subjects randomized, 71, 70, and 74 subjects respectively are included in this summary based on the Full Analysis Set (must have Baseline and at least one post-Baseline efficacy value). This summary uses a Last Observation Carried Forward (LOCF) approach.
Measure: Mean (Standard Deviation); unit: Number of migraine headaches
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Number analyzed (Participants) | 71 | 70 | 74
Number of migraine headaches | -1.4 (3.12) | -1.4 (2.68) | -1.6 (2.10)

2. Secondary Outcome: Change From Baseline in Mean Migraine Headache Rates During the Last 4 Weeks of the Maintenance Period
Time Frame: Baseline, last 4 weeks of the 14-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of migraine headaches
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Number analyzed (Participants) | 71 | 70 | 74
Number of migraine headaches | -1.3 (3.45) | -1.3 (2.82) | -1.7 (2.44)

3. Secondary Outcome: Number of Subjects Who Experience a 50 Percent or Greater Reduction From Baseline in Migraine Frequency During the Entire 14-week Maintenance Period.
Time Frame: Baseline, Entire 14-week Maintenance Period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Number analyzed (Participants) | 71 | 70 | 74
Participants | 26 | 32 | 29

4. Secondary Outcome: Number of Subjects Who Experience a 50 Percent or Greater Reduction From Baseline in Migraine Frequency During the Last 4 Weeks of the Maintenance Period.
Time Frame: Baseline, last 4 weeks of the 14-week Maintenance Period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Number analyzed (Participants) | 71 | 70 | 74
Participants | 27 | 27 | 33

5. Secondary Outcome: Changes From Baseline in Improvement of Function and Reduction of Disability Using the Headache Impact Test (HIT-6)
Description: Headache Impact Test (HIT-6™) consists of 6 items designed to measure the impact headaches have on a person's ability to function. Scores from the 6 questions will be added to create a total score. Range of the total score is 36 to 78. Higher scores indicate a greater impact on the subject's quality of life.
Time Frame: Baseline, last visit in the 17-week Trial Period
Population: Of the 71 (Placebo), 70 (Lacosamide 100mg) and 74 (Lacosamide 300mg) subjects in the Full Analysis Set (must have Baseline and at least one post-Baseline efficacy value), 64, 66, and 66 subjects respectively are included in this summary.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Number analyzed (Participants) | 64 | 66 | 66
Scores on a scale | -3.8 (7.78) | -4.3 (8.67) | -3.5 (8.03)

ADVERSE EVENTS:
Arm/Group | Placebo | Lacosamide 100mg | Lacosamide 300mg
Serious Adverse Events (participants affected / at risk) | 3/72 | 2/72 | 2/74
Other Adverse Events (participants affected / at risk) | 30/72 | 36/72 | 33/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=72) | Lacosamide 100mg (N=72) | Lacosamide 300mg (N=74)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=72) | Lacosamide 100mg (N=72) | Lacosamide 300mg (N=74)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (8) | 4 (5)
Nausea (Gastrointestinal disorders) | 7 (9) | 5 (5) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 5 (5) | 11 (12)
Nasopharyngitis (Infections and infestations) | 7 (7) | 12 (12) | 11 (13)
Influenza (Infections and infestations) | 5 (5) | 3 (3) | 4 (4)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 7 (9) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 4 (6) | 5 (6) | 2 (4)
Headache (Nervous system disorders) | 5 (11) | 3 (9) | 2 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.